CLINICAL TRIAL: NCT04155385
Title: Addiction Treatment Outcome Monitoring Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kevin Hallgren, Associate Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00007996; K01AA024796 (NIH)
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Use Disorder; Substance Use Disorders
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: Non-randomized two-arm clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measurement-only (Active Comparator): Patients will complete weekly measures of treatment progress and goals; however, the information from these measures will not be shared with clinicians or patients.
  Interventions: Other: Measurement
- Measurement and feedback (Experimental): Patients will complete weekly measures of treatment progress and goals; the information from these measures will be shared with clinicians.
  Interventions: Other: Measurement; Other: Feedback

INTERVENTIONS:
Other: Measurement — The measurement system collects information about patients' treatment progress and goals in key areas that are associated with long-term clinical outcomes (e.g., substance use, craving, coping skills, self-efficacy, life satisfaction, depression). Patients complete the measure up to once per week for up to six months.
Other: Feedback — The feedback system is a web-based dashboard that displays current and historical results in each of the outcome and goal domains that is measured; it is available to addiction treatment clinicians who are working with patients enrolled in the study.
  Arms: Measurement and feedback

SUMMARY:
This research evaluates a tool designed for measurement-based care in addiction treatment. Patients in addiction treatment will be invited to complete weekly measures indicating treatment progress and goals. For half the patients, their addiction treatment clinician will be able to view their weekly progress and goals via a secure dashboard. The research will test the feasibility and acceptability of the measurement-based care tool and will evaluate its impact on within-session discussion topics and clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old.
2. Self-reports that they are a patient at Harborview Mental Health and Addiction Services (HMHAS) clinic.
3. Self-reports that they are receiving services at HMHAS clinic for an alcohol or drug-related concern.
4. Has a smartphone with a working phone number and a mobile plan that allows text messages and internet connection.
5. AUDIT-C score indicates past-year hazardous drinking (summed score is at least 3 or 4 for women or men, respectively), or self-reports any drug use for non-medical reasons in the past year.
6. Does not anticipate moving away from the Seattle area within 6 months.
7. Does not anticipate becoming incarcerated in next 6 months.
8. Able to speak and read English (based on self-report).
9. Must be receiving clinical services from an HMHAS clinician who is also participating in the study, which will be evidenced by having at least 3 appointments with a participating HMHAS clinician that were either completed within the past three months or are scheduled to occur within the next three months, verified by the electronic health record.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Measure completion | 6 months
  Logged number of weekly measurement-based care surveys that were completed
Discussion of topics measured by the weekly progress measure | About 6 weeks after enrollment
  Self-reported amount of time spent discussing topics measured in the weekly progress measure. This will be measured via a self-report questionnaire ("In-Session Discussion Topics" questionnaire), which was generated for the current study. The measure will assess the extent to which they discussed each of the following topics in their most recent treatment session: Drinking/drug use, cravings, coping strategies, abstinence self-efficacy, outlook on life, mental health, therapeutic alliance, and treatment goals. Each item is reported on a 4-point Likert scale (minimum value = 0 "did not discuss", maximum value = 3 "discussed extensively" -- higher scores do not necessarily indicate "better" clinical outcomes; however, we hypothesize that the measurement-based care tool will increase the in-session discussion of these topics, and therefore higher outcomes in the measurement-and-feedback group would be consistent with our hypothesis).
Changes in treatment outcomes as measured by the weekly progress measure | 6 months
  Self-reported responses to the weekly progress measure will be evaluated using longitudinal growth curve models. The check-in measure was developed for the current study and consists of items drawn from several existing measures, including the Substance Use Recovery Evaluator, Alcohol Abstinence Self-Efficacy scale, Working Alliance Inventory, and Patient Health Questionnaire-2. The measure is called "The Weekly Check-In" and it provides a "total recovery score" ranging from 0 to 100, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Clinician log-ins to dashboard | 6 months
  Number of log-ins to the clinician-facing dashboard, which will be tracked automatically by the dashboard website.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Hallgren, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hallgren KA, Cohn EB, Ries RK, Atkins DC. Delivering Remote Measurement-Based Care in Community Addiction Treatment: Engagement and Usability Over a 6-Month Clinical Pilot. Front Psychiatry. 2022 Apr 7;13:840409. doi: 10.3389/fpsyt.2022.840409. eCollection 2022. PMID 35463505
- See also: Related Info — https://www.frontiersin.org/articles/10.3389/fpsyt.2022.840409/full

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT04155385/Prot_SAP_000.pdf